CLINICAL TRIAL: NCT06235905
Title: An Open-Label, Single-Group Study to Evaluate the Efficacy and Safety of SPN-820 in Adults With Major Depressive Disorder
Brief Title: Open-Label of SPN-820 in Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Navitor Pharmaceuticals, Inc. (Industry)
Collaborators: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAV-17A-008; SPN-820 (Other: Supernus Pharmaceuticals)
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — NV-5138

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SPN-820 6 x 400 mg capsules (Other)
  Interventions: Drug: NV-5138

INTERVENTIONS:
Drug: NV-5138 — NV-5138 is a novel, orally bioavailable, mechanistic target of rapamycin complex 1 (mTORC1) signaling enhancer
  Other Names: SPN-820

SUMMARY:
This study will evaluate of the efficacy and safety of SPN-820 in Adults With Major Depressive Disorder (MDD)

DETAILED DESCRIPTION:
This is an open-label study of adjunctive SPN-820 (2400 mg) administered orally once every 3 days in adults with MDD

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject, aged 18 to 65 years (inclusive) at screening.
* Diagnosis of MDD according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) for either recurrent or single episode MDD without psychotic features that is confirmed by the Mini International Neuropsychiatric Interview (MINI) at screening.
* MADRS total score of ≥22 for the current major depressive episode (MDE) at screening and baseline (day 1) before study medication (SM) administration.
* CGI-S score of ≥4 (moderately ill or worse) at screening and baseline (day 1) before SM administration.
* Stable, therapeutic dose of one of the following protocol-defined ADTs for the current MDE for ≥6 weeks prior to screening: citalopram, escitalopram, paroxetine, fluoxetine, sertraline, duloxetine, venlafaxine (immediate release or extended release), desvenlafaxine, vilazodone, levomilnacipran, vortioxetine, bupropion, or dextromethorphan/bupropion.
* Stable therapeutic dose of the approved ADT throughout the study.

Exclusion Criteria:

* MADRS total score improvement of ≥25% from the highest to the lowest score from screening to baseline.
* Clinically significant abnormal laboratory profiles, vital sign measurements, or ECGs prior to baseline.
* Lifetime history of psychotic disorder, including but not limited to schizophrenia, MDD with psychotic features, or bipolar I/II disorder with and without psychotic features.
* Diagnosis within the last 12 months before screening or current diagnosis of PTSD, OCD, panic disorder, acute stress disorder, or has a history of intellectual disability, autism, or cluster A or B personality disorder.
* Suicidal behavior or suicidal ideation of type 4 or type 5 based on the C-SSRS in the 1 year before screening; a history of suicide attempt in the last 2 years; or more than 2 lifetime suicide attempts.
* History of substance use disorder within 6 months prior to screening or is currently using or has a positive result (urine drug screen) at screening or baseline for drugs of abuse.
* History of alcohol use disorder within 6 months prior to screening.
* In the investigator's opinion, is unlikely to comply with the protocol or is unsuitable for any other reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-08-18 (Actual); Study Completion 2024-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Viking Clinical Research, Temecula, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SPN-820 (2400 mg): SPN-820 (2400 mg) oral capsules
  Participants received SPN-820 6 x 400 mg capsules administered orally every 3 days for a 7-day treatment period.
Period: Overall Study
Arm/Group | SPN-820 (2400 mg)
Started | 40 (The number of participants reported here is based on the Safety Population which includes all participants who took at least one dose of study medication.)
Completed | 38
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Non-compliant with protocol procedures | 1

BASELINE CHARACTERISTICS:
Population: The number of participants reported here is based on the Safety Population, which includes participants who took at least one dose of study medication.
Arm/Group | SPN-820 (2400 mg)
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (15.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 32
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: Participants]
  United States | 40
MADRS Total Score [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Åsberg Depression Rating Scale is a diagnostic questionnaire used to measure the severity of depressive episodes. It consists of 10 items (reported sadness, apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thoughts) and each question is scored from 0 to 6 for a total score ranging 0 to 60. Higher scores indicate more severe conditions.
  units on a scale | 33.1 (5.41)
HAM-D6 Total Score [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Rating Scale - 6 Items is a diagnostic questionnaire used to measure the severity of depressive episodes. It consists of 6 items (depressed mood, work and activities, somatic symptoms general, feeling of guilt, anxiety psychic, retardation) and each question is scored from 0 to 4 except for one item, somatic symptoms general, which is scored from 0 - 2 for a total score ranging 0 to 22. Higher scores indicate more severe conditions.
  units on a scale | 13.6 (1.69)
CGI-S [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity of Illness is a single-item clinician rating of the clinician's assessment of the severity of symptoms in relation to the clinician's total experience with patients with that condition. CGI-S is evaluated by the Investigator on a 7- point scale with 1=Normal, 2=Borderline ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, and 7=Extremely ill.
  units on a scale | 4.6 (0.64)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Each Time Point in the Hamilton Depression Rating Scale-6 Items (HAM-D6) Total Score (HAM-D6).
Description: The HAM-D6 scale consists of 6 items: five of them (depressed mood, work and activities, feeling of guilt, anxiety, psychic, retardation) are scored on a scale of 0 to 4, and one item (somatic symptoms general) is scored on a scale 0 to 2. The total score is the sum of the 6 items ranging from 0 to 22, higher scores indicate severe depression, and lower scores are better outcomes.
Time Frame: 10 days (end of study)
Population: Full Analysis Set (FAS) Population: the FAS includes all participants who receive at least one dose of study medication and have a baseline and at least one post-baseline measurement of HAM-D6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPN-820 (2400 mg)
Number analyzed (Participants) | 40
score on a scale
  Day 1 - 2 Hours | -6.1 (3.90)
  Day 1 - 4 Hours | -7.2 (3.96)
  Day 1 - 8 Hours | -7.5 (3.59)
  Day 2: number analyzed (Participants) | 39
  Day 2 | -7.8 (3.58)
  Day 3 | -8.7 (3.47)
  Day 4 - Predose: number analyzed (Participants) | 38
  Day 4 - Predose | -7.2 (3.04)
  Day 4 - 2 Hours: number analyzed (Participants) | 38
  Day 4 - 2 Hours | -8.9 (3.45)
  Day 4 - 4 Hours: number analyzed (Participants) | 38
  Day 4 - 4 Hours | -9.5 (3.33)
  Day 4 - 8 Hours: number analyzed (Participants) | 38
  Day 4 - 8 Hours | -9.7 (3.33)
  Day 5: number analyzed (Participants) | 38
  Day 5 | -9.3 (3.37)
  Day 6: number analyzed (Participants) | 37
  Day 6 | -9.8 (3.22)
  Day 7 - Predose: number analyzed (Participants) | 39
  Day 7 - Predose | -9.2 (3.38)
  Day 7 - 2 Hours: number analyzed (Participants) | 39
  Day 7 - 2 Hours | -9.9 (3.09)
  Day 7 - 4 Hours: number analyzed (Participants) | 39
  Day 7 - 4 Hours | -9.7 (3.11)
  Day 7 - 8 Hours: number analyzed (Participants) | 39
  Day 7 - 8 Hours | -10.2 (3.21)
  Day 8: number analyzed (Participants) | 39
  Day 8 | -9.8 (3.15)
  Day 9: number analyzed (Participants) | 38
  Day 9 | -9.9 (2.67)
  Day 10: number analyzed (Participants) | 38
  Day 10 | -9.6 (3.18)

2. Secondary Outcome: Change From Baseline to Each Time Point in the Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score.
Description: MADRS is a 10-item scale (Reported sadness, Apparent sadness, Inner tension, Reduced sleep, Reduced appetite, Concentration difficulties, Lassitude, Inability to feel, Pessimist thoughts, and Suicidal thoughts) where each item is scored from 0 to 6. The total score is the sum of the 10 items ranging from 0 to 60 where higher scores indicate more severe depression, and lower scores are better outcomes.
Time Frame: 10 days (end of study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPN-820 (2400 mg)
Number analyzed (Participants) | 40
score on a scale
  Day 1 - 4 Hours | -16.6 (10.06)
  Day 4 - Predose: number analyzed (Participants) | 38
  Day 4 - Predose | -16.6 (9.05)
  Day 4 - 4 Hours: number analyzed (Participants) | 38
  Day 4 - 4 Hours | -21.2 (9.93)
  Day 7 - Predose: number analyzed (Participants) | 39
  Day 7 - Predose | -21.2 (9.83)
  Day 7 - 4 Hours: number analyzed (Participants) | 39
  Day 7 - 4 Hours | -23.3 (10.60)
  Day 10: number analyzed (Participants) | 38
  Day 10 | -22.9 (9.98)

3. Secondary Outcome: Change From Baseline to Each Time Point in the Clinical Global Impression - Severity of Illness Score (CGI-S).
Description: CGI-S is a single-item clinician rating of the clinician's assessment of the severity of symptoms in relation to the clinician's total experience with patients with that condition. The CGI-I is rated on a 7-point scale from 1 to 7, where 1 = "normal not at all ill" and 7 = "among the most extremely ill patients". Successful therapy is indicated by a lower overall score.
Time Frame: 10 days (end of study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPN-820 (2400 mg)
Number analyzed (Participants) | 40
score on a scale
  Day 4: number analyzed (Participants) | 38
  Day 4 | -1.5 (1.08)
  Day 7: number analyzed (Participants) | 39
  Day 7 | -2.2 (1.21)
  Day 10: number analyzed (Participants) | 38
  Day 10 | -2.4 (1.35)

4. Secondary Outcome: Suicidal Ideation and Behavior as Measured by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS assessment included "yes" or "no" responses for 5 questions, each related to suicidal ideation (wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods, active suicidal ideation with some intent, active suicidal ideation with specific plan) and suicidal behavior (preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, suicide). Number of participants with a response of 'yes' to any suicidal ideation or suicidal behavior item as measured by C-SSRS is reported.
Time Frame: 10 days (end of study)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | SPN-820 (2400 mg)
Number analyzed (Participants) | 40
participants
  Day 1 (Baseline) - Suicidal Ideation | 5
  Day 1 (Baseline) - Behavior | 0
  Day 4 - Suicidal Ideation: number analyzed (Participants) | 39
  Day 4 - Suicidal Ideation | 2
  Day 4 - Suicidal Behavior: number analyzed (Participants) | 39
  Day 4 - Suicidal Behavior | 0
  Day 7 - Suicidal Ideation: number analyzed (Participants) | 39
  Day 7 - Suicidal Ideation | 2
  Day 7 - Suicidal Behavior: number analyzed (Participants) | 39
  Day 7 - Suicidal Behavior | 0
  Day 10 - Suicidal Ideation: number analyzed (Participants) | 39
  Day 10 - Suicidal Ideation | 1
  Day 10 - Suicidal Behavior: number analyzed (Participants) | 38
  Day 10 - Suicidal Behavior | 0

5. Secondary Outcome: Incidence of Treatment Emergent Adverse Events
Description: The incidence of treatment-emergent adverse events (TEAEs) was measured as the percent of participants who took at least one dose of SPN-820 and reported at least one adverse event during 10 days of adjunct treatment. The percent is calculated by dividing "the number of participants who reported at least one Adverse Event" by "the number of participants in the Safety Population" and then multiplying the product by 100. The higher the percent, the higher the incidence.
Time Frame: 10 days (end of study)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | SPN-820 (2400 mg)
Number analyzed (Participants) | 40
percentage of participants | 62.5

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events (TEAEs) were collected after the first dose of study medication up to 12 days (i.e., safety follow up phone call 5 days after the last dose of study medication).
Description: Treatment Emergent Adverse Event (TEAE) is an adverse event (AE) with a start date on or after the first dose of study medication is taken, or that worsened following first administration of study medication.
Arm/Group | SPN-820 (2400 mg)
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 25/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPN-820 (2400 mg) (N=40)
Headache (Nervous system disorders) | 8 (8)
Somnolence (Nervous system disorders) | 6 (8)
Dizziness (Nervous system disorders) | 4 (6)
Cognitive Disorder (Nervous system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (9)
Dry mouth (Gastrointestinal disorders) | 2 (3)
Paraesthesia oral (Gastrointestinal disorders) | 2 (3)
Fatigue (General disorders) | 2 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT06235905/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT06235905/SAP_001.pdf